CLINICAL TRIAL: NCT07400159
Title: Postprandial Thermogenesis in Obese Adolescents: Effect of Weight Loss
Acronym: TEFAL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Emile Roux (Other)
Collaborators: Université Clermont-Auvergne, France (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RIPH2_GADEA_TEFAL; 2025-A01846-43 (Other: ID-RCB)
Record Dates: First submitted 2026-01-20; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Obesity & Overweight
Keywords: dietary thermogenesis in obese adolescents
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adolescents with obesity (Experimental): Adolescents aged 11 to 17 (inclusive), at Tanner stage 3-5 of sexual maturation, With obesity defined as a Quételet index above the 97th percentile according to national curves.
  Interventions: Diagnostic Test: Anthropometric measurements; Diagnostic Test: Body composition assessment; Other: Leeds Foods Preference Questionnaire
- Adolescent with normal weight (Experimental): Adolescents aged 11 to 17 (inclusive) with normal weight
  Interventions: Diagnostic Test: Anthropometric measurements; Diagnostic Test: Body composition assessment; Other: Leeds Foods Preference Questionnaire

INTERVENTIONS:
Diagnostic Test: Anthropometric measurements — For both arms, participants' body weight will be measured to the nearest 0.1 kg using a calibrated manual scale. Height will be measured to the nearest 0.5 cm using a standard wall-mounted height gauge. Waist circumference (WC) will be measured halfway between the last rib and the upper edge of the iliac crest. The Quételet index will be expressed as a Z-score using the "calimco" software adapted to the French population, in order to compare changes in the Quételet index regardless of age and gender.
Diagnostic Test: Body composition assessment — For both arms, body composition will be assessed using dual energy X-ray absorptiometry (DXA, QDR-4500A, Hologic, Inc., Waltham, MA). Scanning the body with an X-ray beam at two different energy levels allows for the measurement of body composition (mineral mass, active tissue mass, and fat mass) and bone geometry in both adults and children. Measurements will be taken of the whole body, the lumbar spine, and the hip, requiring approximately 15 minutes of examination time. This method also involves low radiation exposure (less than a conventional chest X-ray).
  The risks associated with DXA radiation exposure are considered very low (whole body, lumbar spine, and hip) in children aged 10 to 15 (0.0056 mSV).
Other: Leeds Foods Preference Questionnaire — Their relationship with food will be investigated 15 minutes before the test meal and then 1 hour after, using the Leeds Foods Preference Questionnaire developed and validated by the team led by Professor Blundell, a partner in this study. The adolescents will be asked to answer a series of questions about their food preferences by selecting their favorite foods from a selection of images during a 10-minute computer exercise. Similarly, during this exercise, they are asked to use a visual analog scale to estimate how much they would like to eat certain foods presented. Based on their choices and the time taken to respond, the LFPQ assesses the adolescents' degree of "liking" and "wanting." The adolescents must complete this exercise 15 minutes before and after the evening test meal. To avoid any influence on food intake at the next meal, the foods presented during the test are not foods presented during the meal. The objective of this exercise is to assess the response of "liking" and

SUMMARY:
The prevention and management of pediatric obesity require a thorough understanding and consideration of the various components of energy balance (i.e., intake and expenditure) and their interactions. Total energy expenditure (TEE) consists of resting metabolism (RM), energy expenditure induced by physical activity (EEPA), and dietary thermogenesis (DTE). While RM and EEPA are the two main contributors to TEE, DTE is often overlooked, even though it can account for around 10% of our daily energy expenditure. In fact, few studies have prioritized the evaluation of the thermic effect of food (TEF), defined as the increase in energy expenditure above the basal metabolic rate when fasting, despite the fact that it accounts for about 10% of total daily energy expenditure. It has been suggested that TEF may play a role in the development or maintenance of obesity.

Some studies indicate a reduction in TEF in individuals living with obesity, possibly due to lower postprandial activation of the sympathetic nervous system, thereby limiting the thermogenic response after meals. Conversely, several studies have reported no decrease in TEF in individuals living with obesity. Due to these conflicting results, no consensus has been reached on the response of TEF in individuals with obesity compared to those of normal weight.

While our team recently conducted a systematic review of the literature in this area, identifying a glaring lack of evidence, the few results available suggest a potential reduction in TEF in children and adolescents with obesity, contributing to minimizing the optimization of their daily energy balance. In their study, Maffeis and colleagues show, for example, a significantly reduced TEF in adolescents with obesity compared to their normal-weight counterparts, despite a higher-calorie test meal adapted to their energy needs.

These results are consistent with those proposed by Salas-Salvado the following year, which suggest a reduced TEF in obese adolescents, associated with their percentage of body fat.This research suggests the need to consider the effects of weight status, body composition, and the caloric composition of a meal in order to better understand TEF in this population. Furthermore, while our team has repeatedly highlighted adaptations in resting metabolism and exercise metabolism in response to weight loss in obese adolescents, the TEF responses to these interventions have also been little studied in adolescents. To our knowledge, there is only one study that has qualitatively assessed this adaptation of TEF to weight loss in this population. According to the authors, while DHEA was reduced at baseline in obese adolescents compared to their normal-weight counterparts, weight loss appeared to increase DHEA levels, but this remains to be confirmed. In this context, the objective of this study is to evaluate the effects of weight loss on dietary thermogenesis in obese adolescents. It will also compare the thermogenesis of these adolescents before weight loss with that of adolescents of normal weight.

ELIGIBILITY:
Inclusion Criteria: • Adolescents aged 11 to 17 (inclusive), at Tanner stage 3-5 of sexual maturation,

* With obesity defined by a Quételet index above the 97th percentile according to national curves for adolescents with obesity and a Quételet index classifying them as normal weight adolescents for the control group,
* Adolescents affiliated with the social security system or equivalent,
* Adolescent who has been informed and has given written consent to participate in the study.

Exclusion Criteria: • Refusal to participate in the study,

* Refusal of consent by legal guardians,
* Regular consumption of tobacco or alcohol,
* Special diet,
* Participation in regular and intense physical and sporting activities,
* Medical or surgical history deemed by the investigator to be incompatible with the study,
* Presence of diabetes, and any other condition limiting the application of either strategy being tested,
* Adolescents undergoing energy restriction or a weight loss program through physical activity at the time of inclusion or during the last 6 months,
* Taking medication that may interfere with the study results.
* Adolescents with cardiovascular problems, i.e., subjects with a history of cardiovascular and/or neurovascular disease, as well as subjects with cardiovascular and/or neurovascular risk factors (excluding obesity/overweight).
* Surgery in the previous 3 months,
* Adolescents who are currently excluded from another study,
* Pregnant or breastfeeding adolescents,
* Adolescents under guardianship/curatorship or legal protection,
* Parents under guardianship/curatorship or legal protection.

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2026-02-28 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Postprandial energy expenditure (PEE) | 3 months for normal weight adolescents and 6 months for adolescents with obesity

SECONDARY OUTCOMES:
HUNGER SENSATION QUESTIONNAIRE | 3 months for normal weight adolescents and 6 months for adolescents with obesity
  Patients will have to answer 4 questions with answer situated in between "not at all" and "Very much". The questions are: Are you hungry? Do you feel satiated? How much could you eat again? Would you like to eat something?
Leeds Foods Preference Questionnaire | 3 months for normal weight adolescents and 6 months for adolescents with obesity
  Their relationship with food will be investigated 15 min before the test meal and then 1 hour after, using the Leeds Foods Preference Questionnaire. The adolescents will be asked to answer a series of questions about their food preferences by selecting their favorite foods from a selection of images during a 10-min computer exercise. During this exercise, they are asked to use a visual analog scale to estimate how much they would like to eat certain foods presented. Based on their choices and the time taken to respond, the LFPQ assesses the adolescents' degree of "liking" and "wanting." The adolescents will be asked to complete this exercise 15 minutes before and after the evening test meal. To avoid influencing food intake at the next meal, the foods presented during the test are not the same as those presented during the meal. As the aim of this exercise is to assess the response of "liking" and "wanting" to food intake, it is necessary to carry it out before and after the meal.

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratoire AME2P, Université Clermont Auvergne, Aubière, France

IPD SHARING:
Plan to Share IPD: No